CLINICAL TRIAL: NCT03621267
Title: Effects of Interactive Stepping Exercise on Executive Function and Gait Variability in Community-dwelling Older Adults
Brief Title: Interactive Stepping Exercise on Executive Function and Gait Variability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: YM107053F
Record Dates: First submitted 2018-07-29; First posted 2018-08-08 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Health Service for the Aged

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive Stepping Exercise (Experimental): Interactive Stepping Exercise (1 hour, 3 times/week, 12 weeks)
  The 1-hour training program will start with10 minutes warm-up session, after that 40 minutes of ISE, and ended with 10 minutes of cool down session.
  Interactive Stepping Exercise (ISE) will perform on a thin mat that was partitioned into 24 squares. The ISE program included forward, backward, lateral and oblique steps, and step patterns were progressively made more complicated.
  Interventions: Other: Interactive Stepping Exercise
- Home exercise program (Active Comparator): 60 minutes, 3 times/week, 12 weeks of home exercise
  Interventions: Other: Home exercise program

INTERVENTIONS:
Other: Interactive Stepping Exercise — Interactive Stepping Exercise will perform on a thin mat, stepping pattern will display through a monitor screen, immediate auditory feedback will give for adjustment
  Arms: Interactive Stepping Exercise
Other: Home exercise program — Home exercise program includes stretching exercise, general strengthening exercise on lower extremity muscles, posture control and balance exercise.
  Arms: Home exercise program

SUMMARY:
The present study is to examine the effects of interactive stepping exercise on executive function and gait variability in community-dwelling older adults

DETAILED DESCRIPTION:
This is a single blinded, randomized controlled trial. 40 community-dwelling older adults will be recruited and randomly assigned to either experimental group (n=20) or control group (n=20). The 12-week intervention comprises of 1-hour exercise per day and 3 days per week. The experimental group will receive interactive stepping exercise while the control group will be put under home exercise program. Primary outcome measures are executive function and gait variability. Secondary outcome measures include community walking test and other gait parameters (gait velocity, stride length and stride time). The participants will receive assessment at pre- and post-intervention

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling older adults
* age ≥ 65 years old
* able to walk independently outdoor without an assistive device
* Mini-mental state examination ≥ 24
* use an exercise pre-participation health screening form by the American College of Sports Medicine to recruit those participants that are suitable to join the training session

Exclusion Criteria:

* diagnosed of any psychiatric and neurologic disorders such as schizophrenia, stroke, Parkinson, Alzheimer disease, etc.
* any comorbidity or disability that would preclude training

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Trail Making Test | Change from Baseline at 12 weeks
  Executive Function
Stroop Test | Change from Baseline at 12 weeks
  Executive Function
Digit Span Test | Change from Baseline at 12 weeks
  Executive Function
Executive Interview 25 questions | Change from Baseline at 12 weeks
  Executive Function
Gait Variability | Change from Baseline at 12 weeks
  Stride length and Stride time variability

SECONDARY OUTCOMES:
Gait velocity | Change from Baseline at 12 weeks
  Gait speed
Stride length | Change from Baseline at 12 weeks
  The distance covered by the combined step length of each limb during gait
Stride time | Change from Baseline at 12 weeks
  The time elapsed between the first contact of two consecutive footsteps of the same foot
Functional Ambulation in community | Change from Baseline at 12 weeks
  Walk for 400 m distance in community

CONTACTS AND LOCATIONS:
Overall Officials: Yea-Ru Yang, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang-Ming University, Taipei, Beitou, Taiwan